CLINICAL TRIAL: NCT04579744
Title: Postoperative Quality of Life in Surgically Treated Patients With Human Adjuvant Disease: Case Series
Brief Title: Postoperative Quality of Life in Treated Patients With Human Adjuvant Disease
Status: Completed | Type: Observational
Sponsor: Hospital Angeles del Pedregal (Other)
Responsible Party: Principal Investigator, javier lopez, Principal investigator, Plastic and reconstructive surgeon staff, MBA, FACS, Hospital Angeles del Pedregal
Other Study IDs: QoL in HAD
Record Dates: First submitted 2020-09-29; First posted 2020-10-08 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Quality of Life; Granuloma, Foreign-Body
Keywords: human adjuvant disease; quality of life; Reconstructive surgery
MeSH Terms: conditions — Granuloma, Foreign-Body

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: EuroQol 5D questionnaire — EuroQol questionnaire (EQ-5d) facilitates to obtain values of health in the physical, psychological, and social dimensions. It is a standardized non-disease specific instrument to describe and value the health-related quality of life.

SUMMARY:
This study aims to describe the quality of life in patients submitted to surgical excision of the adjuvants and injured surrounding tissue. For this purpose, the EuroQol questionnaire (EQ-5d) facilitates to obtain values of health in the physical, psychological, and social dimensions. It is a standardized non-disease specific instrument to describe and value the health-related quality of life. Although there are only five domains, it has been found to cover the most critical dimensions of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of human adjuvant disease due to foreign substances injection
* Treated surgically to remove foreign substance
* In a private practice setting and treated all by plastic surgeon senior author.

Exclusion Criteria:

* History of antidepressant use during the follow up

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with history of injection of foreign substances as mineral oil or paraffin for cosmetic purposes and who developed human adjuvant disease, characterized for chronic fatigue, myalgias, arthralgias, fever, chronic pain and skin trophic changes due to this foreign substances.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Quality of life: EuroQuality Of Life-5Dimensions | 31.09 months (range 6 - 96)
  Each EuroQOL-5Dimensions instrument comprises a short descriptive system questionnaire and a visual analogue scale (EQ VAS) that are cognitively undemanding, taking only a few minutes to complete. The questionnaire provides a simple descriptive profile of a respondent's health state. Values of health in the physical, psychological, and social dimensions are investigated. After surgical removal of foreign substances quality of life should have high values.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Angeles Pedregal, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Will share info about overall quality of life, also each score of the 5 domains of EQ-5D. Comparison of results with different methods of surgical removal. Share will be in forums, symposia and article sharing